CLINICAL TRIAL: NCT05850832
Title: Efficacy of Esmolol Versus Magnesium Sulphate on Quality of Recovery in Patients Undergoing Laparoscopic Cholecystectomy: Randomized Controlled Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0305810
Record Dates: First submitted 2023-04-29; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Esmolol Adverse Reaction
Keywords: cholecystectomy; recovery profile; opioid sparing
MeSH Terms: interventions — esmolol; Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: 60 patients aged 20-65 years of both sexes, of American society of Anesthesiologists (ASA) physical status I and II planned for ambulatory laparoscopic cholecystectomy under general anaesthesia were engaged to this study.
  * Group (E): (Esmolol group) received loading dose 1 mg/kg followed by maintenance dose of 30 μg/kg/min throughout the surgery.
  * Group (M): (Magnesium sulphate group) received loading dose 40 mg/kg over a period of 15 mins and maintenance 15 mg/kg/h throughout the surgery.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Active Comparator): Esmolol group: patients received loading dose 1 mg/kg followed by maintenance dose of 30 μg/kg/min throughout the surgery
  Interventions: Drug: Esmolol
- Group M (Active Comparator): Magnesium sulphate group: patients received loading dose 40 mg/kg over a period of 15 mins and maintenance 15 mg/kg/h throughout the surgery.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Esmolol — loading dose 1 mg/kg followed by maintenance dose of 30 μg/kg/min throughout the surgery.
  Arms: Group E
Drug: Magnesium sulfate — loading dose 40 mg/kg over a period of 15 mins and maintenance 15 mg/kg/h throughout the surgery.
  Arms: Group M

SUMMARY:
sixty patients, of both sexes, of ASA I or II planned for ambulatory laparoscopic cholecystectomy under general anaesthesia were engaged into 2 groups. Esmolol group were given 1 mg/kg loading dose followed by 30 μg/kg/min throughout the surgery, whereas magnesium sulphate (MgSo4) group were given loading dose 40 mg/kg over 15 mins then maintenance dose 15 mg/kg/h till end of surgery. General anaesthesia was standardized and postoperative analgesia included fentanyl. Variables denoting immediate recovery from anaesthesia, pain score and time of stay in PACU were recorded. White-Song score ≥ 12 along with pain score < 4 were the cut off levels for patients' discharge from PACU.

DETAILED DESCRIPTION:
The primary end point of this study are variables concerning immediate postoperative recovery like times needed for spontaneous eye opening, tongue protrusion, extubation and ability of the patient to mention name. Secondary outcomes includes pain assessment using pain numerical scale, time for first call to analgesia, total amount of intraoperative fentanyl consumption, total dose of rescue antiemetics and time of discharge from PACU.

Following attaining Ethical committee approval and patient's written consent- after broad explanation of the entire procedure- 60 patients aged 20-65 years of both sexes, of American society of Anesthesiologists (ASA) physical status I and II planned for ambulatory laparoscopic cholecystectomy under general anaesthesia were engaged to this study.

Exclusion criteria were: patients on chronic use or known allergic to the study drugs, body mass index >35 kg/m2, significant organ dysfunction, cardiac dysrhythmias, neuromuscular diseases, liver or renal disease, known asthma or reactive airway diseases.

Preoperatively all participants were carefully evaluated via detailed history taking, thorough physical examination and routine investigations (complete blood picture, renal function tests and liver functions). Also, they were instructed in the utilization of the verbal rating scale (VRS).

For blinding purpose, both the study drugs were prepared by an anaesthesiologist not enrolled in data assumption. Accordingly, for every case 2 prefilled syringes; one 10-ml for loading dose and the other 20-ml for maintenance infusion were given unidentified to the operating theater containing either Esmolol (Esmolol hydrochloride; Baxter Healthcare Corp., Deerfield, USA) or MgSo4 ( Egyptian international pharmaceutical indust., EYGPT).

Randomization was achieved prior to the study by means of randomization table prepared by computer software to assign the number of cases among the studied groups. Patients were randomly allocated using closed envelopes method into 2 equal groups (n=30 each):

* Group (E): (Esmolol group) received loading dose 1 mg/kg followed by maintenance dose of 30 μg/kg/min throughout the surgery.
* Group (M): (Magnesium sulphate group) received loading dose 40 mg/kg over a period of 15 mins and maintenance 15 mg/kg/h throughout the surgery.

Loading dose was given after fentanyl injection and before propofol induction. Maintenance dose was continued until the end of the procedure.

No premedication was offered. On arrival to the operating room, an intravenous cannula was placed and secured before induction of anaesthesia and all patients were attached to standard monitors including pulse oximetry, ECG, non- invasive blood pressure and end tidal carbon dioxide (ETCO2) monitor (Datex ohmeda S/5).

Anaesthesia was induced with 1 μg/kg fentanyl and 1.5 - 2 mg/kg propofol till cessation of verbal contact. Cisatracurium 0.15 mg/kg was used for neuromuscular relaxation and endotracheal intubation (via 8 or 8.5 mm for males, 7 or 7.5 mm for female patients, high-volume/low pressure portex endotracheal tubes). Soon after induction, in both groups IV dexamethasone 8 mg was given and 1 g paracetamol IV was infused over 15 mins. Anaesthesia was maintained with sevoflurane 1-2 % with 50 % oxygen in air. Increments of IV fentanyl 0.5 µg/kg was given for analgesia if systolic blood pressure or heart rate was increased by more than 20 % of baseline level, also incremental dose of cisatracurium 0.03 mg/kg was used to maintain muscle relaxation according to nerve stimulation. Patients were mechanically ventilated to maintain ETCO2 between 33-35 mmHg and an oxygen saturation of 98 %. The port sites were infiltrated by the surgical team with 3ml of 0.25% bupivacaine. Pneumoperitoneum with carbon dioxide was achieved, maintaining the intraabdominal pressure at 12 mm Hg throughout surgery. Patients were positioned in 30 degrees anti-Trendelenburg position and rotated toward the left side to facilitate exposure of the gall bladder. IV warmed 0.9 % NaCL was given during surgery at a rate 6 ml/kg/hr. If required, intraoperative hypotension (mean arterial blood pressure lower than 50 mm Hg) and bradycardia (heart rate < 40 bpm) were managed in both groups with i.v ephedrine and atropine respectively. At the end of surgery, patients were returned to the supine position and the Co2 left in the peritoneal cavity was expelled by abdominal compression slowly. 0.25 % bupivacaine was injected again at the surgical incisions. Esmolol and Mgso4 infusions were stopped and discarded at end of the procedure, which was marked at the end of skin closure and wound coverage. Anaesthesia was discontinued and 100 % oxygen was administrated. Reversal of muscle relaxants by i.v neostigmine 0.04-0.08 mg/kg and atropine 0.02 mg/kg, and then oral secretion was suctioned and the patients were extubated fully awake after return of the protective airway reflexes with full muscle power. Times passed from end of procedure till spontaneous eye opening (from cessation of infusions till spontaneous eye opening), extubation, tongue protrusion, and patient's ability to mention name were recorded. Duration of surgery (time from skin incision till end of procedure) and duration of anaesthesia (time from induction till shifting the patients from operating table to the PACU) were also recorded.

Patients were transferred to the postanesthesia care unit (PACU) where heart rate, arterial blood pressure, respiration, and temperature were continuously monitored by a nurse blind to the study deign to avoid bias. Postoperative pain management included 1 g of paracetamol IV at 8 hr. Assessed of postoperative pain was done using pain numerical rating scale (NRS) on immediate arrival to PACU and every 30 mins for the first 2 hours afterwards. NRS is a (0-10) scale, where (0) denotes no pain, whereas (10) refers to maximal pain imagined. Fentanyl (25 μg) IV was used when NRS exceeded 4. Times to first rescue analgesia and total amount of fentanyl consumed were recorded. Recue antiemetic ondansetron (4 mg) IV was given for nausea lasting > 5 min (persistent) or vomiting and repeated as required. Total dose of ondansetron was noted.

The White-song scoring system a more up to date quick track scoring framework incorporating fundamental fast track variables like physical steadiness, vitals and consciousness level has been proposed to evaluate the recovery profile. Furthermore it involved assessment of adverse events like postoperative pain and vomiting, which were unfortunately missed by the modified Aldrete score. A minimum score (12 / 14) should be established prior to patient safe fast-tracked. It was evaluated on immediate arrival to PACU and every 30 mins for the first 2 hours afterwards. Patients reached White-Song score 12 + NRS < 4 were discharged from PACU. Length of stay in PACU till discharge were also recorded

ELIGIBILITY:
Inclusion Criteria:

* patients aged 20-65 years of both sexes

Exclusion Criteria:

* patients on chronic use or known allergic to the study drugs
* body mass index >35 kg/m2,
* significant organ dysfunction, cardiac dysrhythmias, neuromuscular diseases
* liver or renal disease,
* known asthma or reactive airway diseases.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
times needed for spontaneous eye opening | immediately postoperative
  time passed from end of procedure until the patient open his eyes

SECONDARY OUTCOMES:
total amount of intraoperative fentanyl consumption | immediately postoperative
  total amount of intra-opertaive fentanyl consumed throughout the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicin, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No